CLINICAL TRIAL: NCT06363136
Title: Evaluation of Foot Posture, Muscle Strength, Functional Performance, and Postural Control in Children With Isolated Gastrocnemius Tightness
Brief Title: Foot Posture, Strength, Performance, and Postural Control in Isolated Gastrocnemius Tightness
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Deniz Tuncer, Assistant professor, Bezmialem Vakif University
Other Study IDs: 14.06.2023-111176
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Gastrocnemius Tightness; Postural Control; Muscle Strength; Functional Performance; Foot Posture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: The group will include 14 children aged 7-16 who are voluntarily participating and being followed for bilateral isolated gastrocnemius tightness by the Department of Orthopedics and Traumatology at Bezmialem Vakif University.
- Control group: The group will consist 14 healthy children from the same age group.

SUMMARY:
Studies on gastrocnemius tightness in healthy children are limited, but there is evidence that ankle dorsiflexion decreases with increasing age in children. It is not known whether gastrocnemius tightness is a normal finding in children, but recurrent leg pain is common in children. It is also known that flexible flatfoot is a normal observation in developing children and that the medial longitudinal arch develops during the first decade of life. Both foot morphology and ankle dorsiflexion change in developing children; however, it is not known whether there is a relationship between them or not.

In the literature, there is no study evaluating foot posture, muscle strength, functional performance, and postural control in children with isolated gastrocnemius muscle tightness. It was planned to evaluate postural control using computerized dynamic posturography (Biodex Balance System), lower extremity muscle strength using a hand-held dynamometer, foot posture using the Foot Posture Index (FPI-6), and functional performance using single-foot-double-foot jump tests in healthy children with isolated gastrocnemius muscle tightness.

DETAILED DESCRIPTION:
Since the gastrocnemius muscle spans both joints, the kinematics of the ankle joint are influenced by knee flexion. According to Kendall & McCreary's assessment of normal joint motion angles, when the knee joint is in extension, the passive dorsiflexion angle of the ankle is approximately 20°, and with knee flexion, the angle can approach 30° due to the relaxation of the gastrocnemius. During the midstance phase of walking, the ankle joint allows for 8-10° of dorsiflexion movement. The evaluation of gastrocnemius muscle tightness is conducted using the Silfverskiold method. However, there are variations in the definitions proposed for the detection of isolated gastrocnemius tightness. In our investigation, when ankle dorsiflexion rises by at least 10° more in knee flexion than knee extension, isolated gastrocnemius tightness will be taken into account.

Isolated gastrocnemius tightness during walking can result in compensatory effects on the lower extremity and foot, causing biomechanical changes such as pes planus, talus eversion, rearfoot pronation, and various symptoms such as plantar fasciitis, leg pain, metatarsalgia, and Achilles tendinopathy. The association between increased rearfoot pronation and isolated gastrocnemius tightness has been demonstrated in the literature. Regardless of the etiology of rearfoot pronation, adaptive isolated gastrocnemius shortening will occur in conjunction with talar plantar flexion. Isolated gastrocnemius tightness causing plantar flexion at the ankle joint and pronation at the subtalar joint also hinders the normal distribution of load on the plantar surface during weight-bearing. Reviewing the literature, it is observed that the effects of isolated gastrocnemius tightness on foot posture, functional parameters, and gait dynamics, especially rearfoot pronation, are reported.

Studies on gastrocnemius tightness in healthy children are limited, but there is evidence that ankle dorsiflexion decreases with age in children. While it is unknown whether gastrocnemius shortening is a normal finding in children, recurrent leg pain is common in children. Additionally, flexible flatfoot is considered a normal observation in developing children, and it is known that the medial longitudinal arch develops in the first ten years of life. Both foot morphology and ankle dorsiflexion change in developing children, but it is unknown whether there is a relationship between the two.

In the literature, there is no study evaluating foot posture, muscle strength, functional performance, and postural control in children with isolated gastrocnemius muscle shortening. In our study, we plan to assess postural control using computerized dynamic posturography (Biodex Balance System), lower extremity muscle strength using a hand-held dynamometer, foot posture using the Foot Posture Index (FPI-6), and functional performance using single-leg and double-leg hop tests in healthy children with isolated gastrocnemius muscle shortening.

ELIGIBILITY:
Inclusion Criteria:

Study group

* Presence of bilateral isolated gastrocnemius tightness (The test is considered positive when ankle dorsal flexion dorsiflexion increases over a minimum of 10 degrees with the knee flexed than the knee extension.
* Being between 7-16 years of age
* Body mass index within normal limits (18.5-24.9 kg/m2) Exclusion criteria
* Presence of high femoral anteversion, internal tibial torsion, and metatarsus adductus
* Presence of hypermobility (Beighton score >4 and above)
* Leg length discrepancy
* Presence of any neurological, rheumatic, musculoskeletal, metabolic, and connective tissue disease
* History of pain, deformity, or surgery associated with the vertebral column and lower extremities
* Presence of cognitive, mental, and/or severe psychiatric illness
* Participation in any exercise program or sportive activity in the last six months

For the control group, the same inclusion/exclusion criteria will be accepted except that the bilateral Silfverskiold test is negative.

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will recruit 14 children aged 7-16 years who were followed up by Bezmialem Vakıf University Department of Orthopaedics and Traumatology for bilateral isolated gastrocnemius tightness who participated voluntarily. In addition, 14 healthy children of the same age group consisting of relatives of the participating families and healthy relatives of the students studying in the department will be included. The cross-sectional study will be conducted in accordance with the Declaration of Helsinki.
  After obtaining informed consent from both parents and children, all evaluations and tests for the participants will be performed at Bezmialem Vakıf University Faculty of Health Sciences Paediatric and Cardiac Physiotherapy and Rehabilitation Education and Research Laboratories.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Postural Control Assessment | 1 day
  Postural stability, limits of stability, and sensory integration of balance will be assessed using the Biodex Balance System®.
Lower extremity muscle strength measurement | 1 day
  The strength of hip adductors-abductors, external-internal rotators, flexors-extensors, knee flexors-extensors, and ankle dorsiflexors-plantar flexors, invertors-evertors muscles will be evaluated isometrically using a handheld dynamometer (MicroFET 2 force gauge, Hoggan Health Industries, Salt Lake City, Utah).

SECONDARY OUTCOMES:
Foot posture assessment | 1 day
  The Foot Posture Index (FPI-6) will be used to assess foot alignment in different planes. Six analyses will be scored on a +2 to -2 scale, and the total score will be recorded.
Functional performance assessment | 1 day
  The Single Leg and Double Leg Horizontal Jump Testswill be used to evaluate lower extremity functional performance.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Tuncer, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eren-Zengin F, Tuncer D, Senaran H, Uzer G. Effects of isolated gastrocnemius tightness on foot posture, strength, function, and balance in children aged 7-16: a case-control study. BMC Sports Sci Med Rehabil. 2025 Oct 3;17(1):289. doi: 10.1186/s13102-025-01210-6. PMID 41039620